CLINICAL TRIAL: NCT04149821
Title: Phase II Study of Umbralisib Plus Ublituximab (U2) in Progressive CLL After Novel Therapy
Brief Title: Umbralisib Plus Ublituximab (U2) in Progressive CLL After Novel Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to low accrual
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-06020316
Record Dates: First submitted 2019-10-30; First posted 2019-11-04 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Chronic Lymphocytic Leukemia; CLL Progression; CLL/SLL
Keywords: CLL; progression
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Disease Progression | interventions — umbralisib; ublituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A Post BTKi Therapy (Experimental): Patients who progress after a BTKi containing regimen
  Interventions: Drug: Umbralisib; Drug: Ublituximab
- Cohort B Post BCL-2 Therapy (Experimental): * Patients who progress after BCL-2 containing regimens
  * Patients who progress on a regimen containing both a BTKi and a BCL-2 inhibitor
  Interventions: Drug: Umbralisib; Drug: Ublituximab

INTERVENTIONS:
Drug: Umbralisib — * Lead-in cycle of 28 days (Cycle -1) of umbralisib monotherapy, 800mg oral daily
  * Continued 800mg oral daily dosing in all subsequent cycles (combination therapy cycles 1-6, then continued monotherapy cycle 7 and beyond)
  Other Names: TGR-1202
Drug: Ublituximab — -Co-administered on days 1 and 2 (dose split over days 1 and 2), 8, 15 of cycle 1 then on day 1 for subsequent cycles 2-6
  Other Names: TG-1101

SUMMARY:
This study evaluates the efficacy and safety of umbralisib and ublituximab (U2) as salvage therapy in patients with chronic lymphocytic leukemia (CLL) who have progressed either on a BTK inhibitor (BTKi) or BCL-2 inhibitor. The study will evaluate this combination in two parallel cohorts and subjects will be assigned based on which class of novel agent-containing regimen was used prior. Cohort A will consist of patients who progress after BTKi containing regimens and Cohort B will consist of patients who progress after a BCL-2 containing regimen. Subjects who progress on a regimen containing both a BTKi and a BCL-2 inhibitor, will be enrolled in cohort B. Each cohort will be evaluated independently of each other.

DETAILED DESCRIPTION:
This is a single-center, two cohort Phase 2 clinical trial investigating the effectiveness of umbralisib and ublituximab in patients with progressive CLL. Cohort A will consist of patients who who have progressed after receiving either a BTK inhibitor (BTKi) or BCL-2 inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of CLL based upon 2018 International Workshop on CLL (IWCLL) criteria.
* Patient must have progressed on a BTK or BCL-2 containing regimen as the prior line of therapy. Patients who were treated with a regimen containing both classes of novel agents will be allowed to enroll and will be enrolled into Cohort B. Patients who receive a temporizing non-experimental treatment such as an anti-CD20 monoclonal antibody, corticosteroid including high dose methylprednisolone after progression on a BTK or BCL-2 inhibitor will be considered for enrollment after discussion with the study sponsor.
* Age ≥18 years
* ECOG performance status ≤2
* Patient must have adequate bone marrow function and meet the below thresholds:

  * Absolute neutrophil count of ≥ 750 cell/μL in absence of G-CSF for 7 days prior to enrollment.
  * Platelet count of ≥ 30,000 cells/μL, or ≥ 20,000 cells/μL if there is bone marrow involvement)
* Patient must have adequate organ function and meet the thresholds below:

  * Total bilirubin ≤ 1.5 times the upper limit of normal (ULN). Subjects with bilirubin exceeding this limit due to Gilbert's disease are eligible
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 x ULN if no liver involvement or ≤5 x the ULN if known liver involvement
  * Creatinine clearance >30 ml/min/1.73m2 as calculated by the MDRD equation
* Ability to swallow and retain oral medication.
* Females who are not of child-bearing potential, and females of child-bearing potential (FCBP) who have a negative serum pregnancy test within 3 days prior to initial trial treatment. Males of reproductive potential may not participate unless they agree to use medically acceptable contraception. FCBP and all male partners, and male subjects must consent to use a medically acceptable method of contraception throughout the study period and for 4 months after the last dose of study drug
* Willingness and ability to comply with trial and follow-up procedures, and give written informed consent

Exclusion Criteria:

* Patient has had prior exposure to a PI3K inhibitor at any point in treatment history
* Patient has discontinued the BTK or BCL2 inhibitor due to intolerance. Intolerance will be defined as discontinuing prior BTKi or BCL-2 therapy for any reason without evidence of progression. Patients who were re-challenged after discontinuation for therapeutic reasons will be allowed if the toxicity did not recur or was managed without indication for discontinuation. Patients who progress on BTKi or BCL-2 therapy who were on a reduced dose due to an AE/intolerance are eligible as long as progression has been documented on that reduced dose.
* Patient has clinical or radiographic evidence of, or has biopsy proven Richter's transformation or prolymphocytic leukemia.
* Patient has undergone an allogeneic stem cell transplant.
* Patient has received an autologous hematologic stem cell transplant within 6 months of study entry.
* Prior history of malignancy within 3 years of study enrollment except for adequately treated basal, squamous cell carcinoma or non-melanomatous skin cancer, carcinoma in situ of the cervix, superficial bladder cancer not treated with intravesical chemotherapy or BCG within 6 months, localized prostate cancer and PSA <1.0 mg/dL on 2 consecutive measurements at least 3 months apart with the most recent one being within 4 weeks of study entry.
* Patient is known to be positive for HIV.
* Patient has history of hepatitis C infection, active infection with hepatitis B or active cytomegalovirus (CMV) as determined by PCR.
* Patient has previous exposure to a BTK inhibitor therapy within 14 days of initiating study treatment on Cycle 1 Day 1, or previous exposure to anti-cancer therapy including chemotherapy, radiotherapy, or investigational therapy, including other targeted small molecule agents within 21 days of initiating study treatment on Cycle 1 Day 1.
* Evidence of ongoing systemic bacterial, fungal or viral infection, except localized fungal infections of skin or nails.
* History of anaphylaxis (excluding infusion related reactions) in association with previous anti-CD20 administration.
* Inflammatory bowel disease (such as Crohn's disease or ulcerative colitis).
* Malabsorption syndromes.
* Irritable bowel syndrome with greater than 3 loose stools per day as a baseline.
* Any severe and/or uncontrolled medical conditions or other conditions that could affect participation in the study such as:

  * Symptomatic, or history of documented congestive heart failure (New York Heart Association functional classification III-IV)[see Appendix: NYHA Classifications]
  * Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, CHF, or myocardial infarction within 6 months of enrollment.
  * Concomitant use of medication known to cause QT prolongation or torsades de pointes should be used with caution and at investigator discretion.
  * Poorly controlled or clinically significant atherosclerotic vascular disease including cerebrovascular accident (CVA), transient ischemic attack (TIA), angioplasty, cardiac or vascular stenting within 6 months of enrollment.
* Females who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Allan, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: WCM Joint Clinical Trials Office — https://jcto.weill.cornell.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A Post BTKi Therapy: Patients who progress after a BTKi containing regimen
  Umbralisib: -Lead-in cycle of 28 days (Cycle -1) of umbralisib monotherapy, 800mg oral daily
  -Continued 800mg oral daily dosing in all subsequent cycles (combination therapy cycles 1-6, then continued monotherapy cycle 7 and beyond)
  Ublituximab: -Co-administered on days 1 and 2 (dose split over days 1 and 2), 8, 15 of cycle 1 then on day 1 for subsequent cycles 2-6
- Cohort B Post BCL-2 Therapy: * Patients who progress after BCL-2 containing regimens
  * Patients who progress on a regimen containing both a BTKi and a BCL-2 inhibitor
  Umbralisib: -Lead-in cycle of 28 days (Cycle -1) of umbralisib monotherapy, 800mg oral daily
  -Continued 800mg oral daily dosing in all subsequent cycles (combination therapy cycles 1-6, then continued monotherapy cycle 7 and beyond)
  Ublituximab: -Co-administered on days 1 and 2 (dose split over days 1 and 2), 8, 15 of cycle 1 then on day 1 for subsequent cycles 2-6
Period: Overall Study
Arm/Group | Cohort A Post BTKi Therapy | Cohort B Post BCL-2 Therapy
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 0 subjects were enrolled in Cohort A.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A Post BTKi Therapy | Cohort B Post BCL-2 Therapy | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 1 | 1
  >=65 years |  | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 | 1
  Male |  | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 1 | 1
  Not Hispanic or Latino |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 0 | 0
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Umbralisib in Combination With Ublituximab (U2) as Measured by Overall Response Rate (ORR) in Patients With CLL Who Have Progressed on a BTKi or BCL-2 Inhibitor
Description: Number of subjects who achieve a partial or complete response
Time Frame: 11 months
Population: 0 subjects were enrolled in Cohort A.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A Post BTKi Therapy | Cohort B Post BCL-2 Therapy
Number analyzed (Participants) | 0 | 1
Participants |  | 0

2. Secondary Outcome: Safety of Umbralisib in Combination With Ublituximab (U2) as Measured by the Percentage of Subjects Who Experience 1 or More Adverse Events
Description: Rate of subjects who experience 1 or more adverse events
Time Frame: 1 year and 4 months
Population: 0 subjects were enrolled in Cohort A.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A Post BTKi Therapy | Cohort B Post BCL-2 Therapy
Number analyzed (Participants) | 0 | 1
Participants |  | 1

3. Secondary Outcome: Complete Remission Rate as Measured by the Number of Subjects Who Achieve Complete Response as Their Best Response
Description: Number of subjects who achieve complete response on study
Time Frame: 1 year and 4 months
Population: 0 subjects were enrolled in Cohort A.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A Post BTKi Therapy | Cohort B Post BCL-2 Therapy
Number analyzed (Participants) | 0 | 1
Participants |  | 0

4. Secondary Outcome: Duration of Response
Description: Median interval of time between subjects' first objective response to the first sign of disease progression
Time Frame: 1 year and 4 months
Population: 0 subjects were enrolled in Cohort A.
Measure: Number; unit: years
Arm/Group | Cohort A Post BTKi Therapy | Cohort B Post BCL-2 Therapy
Number analyzed (Participants) | 0 | 1
years |  | 0

ADVERSE EVENTS:
Time Frame: 1 year and 3 months
Description: 0 subjects were enrolled in Cohort A."
Arm/Group | Cohort A Post BTKi Therapy | Cohort B Post BCL-2 Therapy
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/1
Other Adverse Events (participants affected / at risk) | 0/0 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A Post BTKi Therapy (N=0) | Cohort B Post BCL-2 Therapy (N=1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 3
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Grade 3
Syncope (Nervous system disorders) | 0 (0) | 1 (1) — Grade 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A Post BTKi Therapy (N=0) | Cohort B Post BCL-2 Therapy (N=1)
Blurred vision (Eye disorders) | 0 (0) | 1 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (5)
Headache (Nervous system disorders) | 0 (0) | 1 (7)
Fatigue (General disorders) | 0 (0) | 1 (13)
Lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (6)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (7)
Hypocalcemia (Investigations) | 0 (0) | 1 (2)
Creatinine increased (Investigations) | 0 (0) | 1 (3)
Thrombocytopenia (Investigations) | 0 (0) | 1 (5)
Dysuria (Hepatobiliary disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tongue numbness (General disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Numbness (General disorders) | 0 (0) | 1 (2)
Neuropathy (Nervous system disorders) | 0 (0) | 1 (3)
Axillary Lymphadenopathy (General disorders) | 0 (0) | 1 (2)
Abdominal Pain (General disorders) | 0 (0) | 1 (2)
Constipation (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (2)
Mouth Sores (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study did not reach the target number of participants needed to achieve target power and statistically reliable results

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/21/NCT04149821/Prot_SAP_000.pdf